CLINICAL TRIAL: NCT07280169
Title: Identifying Non-Union Rates Using Carbo-fix Lateral Plate Devices and Standard Plate-Nail Construct in Distal Femur Fractures
Brief Title: Carbo-fix Lateral Plate Devices and Standard Plate-Nail Constructs in Distal Femur Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: CarboFix Orthopedics Ltd. (Industry)
Responsible Party: Principal Investigator, Kyle Schweser MD, ASSOCIATE PROFESSOR OF ORTHOPAEDIC SURGERY, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2097810
Record Dates: First submitted 2025-11-20; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Distal Femur Fracture
Keywords: Distal Femur Fracture; Carbofix; Plate-Nail Construct
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Carbo-fix Lateral Plate Device (Active Comparator)
  Interventions: Device: Carbo-fix Lateral Plate Device
- Standard Plate-Nail Construct (Active Comparator)
  Interventions: Device: Standard Plate-Nail Construct

INTERVENTIONS:
Device: Carbo-fix Lateral Plate Device — Participants that are randomized to this group will have their distal femur fracture repaired with the Carbofix carbon fiber lateral locking plate
  Arms: Carbo-fix Lateral Plate Device
Device: Standard Plate-Nail Construct — Participants who randomize to this group will have their distal femur fracture repaired with the standard lateral plate and intramedullary nail construct.
  Arms: Standard Plate-Nail Construct

SUMMARY:
The purpose of this randomized clinical trial is to decrease non-union rates in distal femur fracture fixation. Carbo-fix lateral femur plate and standard intramedullary nail-plate constructs have been shown to have lower non-union rates. With decreased non-union rates, re-operation rates will decrease, leading to improved patient outcomes and clinical care. This study will randomize patients to one of the two groups. Then investigators will be collecting data on the standard plate and nail combination and compare outcomes with the Carbofix plate to see differences in union rates. All procedures are currently standard of care and no procedures are research only.

DETAILED DESCRIPTION:
Distal femur fractures are quite common, accounting for 3-6% of all femur fractures. In young adults, high energy trauma is most likely the cause, whereas in the elderly population, a low energy trauma due to osteoporosis is likely. Mortality for elderly patients with distal femur fractures is <20% at 1 year and approximately 50% at 5 years. Standard of care treatment for distal femur fractures is open reduction and internal fixation with locking plates, condylar screws, blade plates, or intramedullary nails, depending on the fracture characteristics. Non-union is a known complication of distal femur fixation; recent studies have shown non-union rates up to 33% with lateral locking plating. Patient factors and fracture patterns contribute significantly to the observed success of distal femur fixation operations.

A combined nail-plate fixation has increased in use in recent years, aiming to improve stability and allow early weightbearing. The nail-plate combination significantly increases the chances of the union and is generally used in non-union cases. Its use has flourished and is now an option for primary repair of distal femur fractures. Garala et al compared outcomes among fixation with a single lateral plate and a combined nail-plate construct and found 11 non-unions within the single lateral plate group compared to none in the nail-plate construct.

Metal plates and nails are commonly used for fixation. Carbon fiber, an emerging modality in orthopaedic surgery, has unique physical, chemical, and biological characteristics. It has a high strength to weight ratio and greater tensile strength compared to metallic materials, 7.5 times that of aluminum and 4 times that of steel. A retrospective study using carbon fiber lateral plates in supracondylar periprosthetic femur fractures in elderly patients reported all fractures resulting in union. When compared to titanium, carbon fiber had increased strength, stiffness, and lower wear resistance, as well as an elastic modulus half of bone. The Carbo-fix nails made of CF-PEEK have an advantage relative to metallic nails, although features are similar. These nails offer advantages related to imaging, as they are radiolucent on fluoroscopy and normal radiograph and decrease artifact on CT and MRI.

The purpose of this randomized clinical trial is to decrease non-union rates is distal femur fracture fixation. Carbo-fix lateral femur plate and standard intramedullary nail-plate constructs have been shown to have lower non-union rates. With decreased non-union rates, re-operation rates will decrease, leading to improved patient outcomes and clinical care. This study will be collecting data on the standard plate and nail combination and compare outcomes with the Carbofix plate to see differences in union rates. All procedures are currently standard of care and no procedures are research only.

Lateral plates and intramedullary nails are used as standard of care for distal femur fractures. Metal plates and nails are typically used, but the Carbofix carbon fiber version of the lateral locking plate can be used as standard of care as well. Non-union rates in the metal lateral locking plates are 20-33%, whereas the carbon fiber plates have a 3-9% non-union rate. The nail-plate combination has a 1-3% non-union rate. Using the Carbofix carbon fiber lateral plates and the standard nail-plate combination can reduce non-union rates in patients and provide better outcomes.

The investigators will be investigating the Carbofix carbon fiber lateral locking plate in this study due to its low non-union rate. This plate is used for distal femur fracture fixation and is FDA approved. Subjects will be randomized to receive the Carbofix carbon fiber lateral locking plate or the typical metal lateral plate and nail combination.

The University of Missouri typically uses the standard metal lateral locking plate and intramedullary nail to treat distal femur fractures. Both are FDA approved.

Study candidates will be screened and identified at morning trauma conference and on the trauma surgery schedule at the University of Missouri Hospital and at Missouri Orthopaedic Institute. A member of the research team will interview the patient in their room while they are at the University of Missouri Hospital/Missouri Orthopaedic Institute. The study, protocol, and consent will be explained to the patient. The patient is encouraged to ask questions and demonstrate understanding of the study. After this, the investigators will obtain informed consent per the IRB protocol. Each candidate will receive a copy of the consent to review with family. Members of the clinic team and research team will collect patient information, previous surgery history, and demographics, including age, sex, BMI, smoking status, and other co-morbidities. This will be collected from the electronic medical chart as well as the patient interview.

The investigators anticipate enrolling 50 patients in the carbon fiber lateral plate cohort and 50 patients in the standard lateral plate plus nail combination cohort over a 2-year enrollment period.

Eligible candidates will be enrolled into the study prior to surgery. Patients will be asked if pregnant. Once informed consent is obtained, the research team will randomize the participant to the carbon fiber lateral plate only or the standard plate-nail combination, both standard of care procedures. A sealed envelope with plate only or plate and nail combination will be opened by a member of the research team. The surgeon will be made aware of which construct will be used prior to surgery. The surgeon will discuss the treatment arm and explain risks to the patient.

Surgical information will be recorded, including length of surgery (in minutes), blood loss, complications during surgery, and any antibiotics used during surgery. Pain medication used following surgery, length of stay, and changes in discharge will also be recorded.

Patients will follow up at standard of care visits - 2 weeks, 6 weeks, 3 months, 6 months, 1 year. At each visit, patients will answer PROs and receive x-rays as per standard of care. Radiographs will be assessed for union; once union is achieved, time to union will be recorded. Pain and pain medication use will be recorded at each subsequent visit. PROs include VAS pain score, PROMIS physical function, and PROMIS pain interference will be recorded as well.

There is minimal risk with breach of confidential medical information. Efforts will be made to avoid the breach of confidentiality. Records are given a study identification number that will be free of subject's name and identifiers. Identification numbers connected with subjects' names will be kept in a secure location and otherwise will be archived in a secure storage facility or destroyed.

Anticipated benefits include possible reduction in non-union rates, which could lead to better patient outcomes and improved treatment in orthopaedic surgery.

Subject safety will be ensured through standard of care procedures and monitoring by clinical and surgical staff.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years or older, with a distal femur fracture requiring surgery
* Adult patients able to understand and sign the consent and answer PROs

Exclusion Criteria:

* Age under 18 years
* Currently pregnant or breastfeeding (patient will simply be asked pregnancy status)
* Unable to give consent
* Prisoner
* Mentally disabled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
The total number of participants that have non-union of their distal femur fractures when utilizing a carbon fiber lateral plate only or a standard nail/plate combination as assessed by standard of care radiographs. | 1 year

SECONDARY OUTCOMES:
The average scores of the patient reported outcomes for pain scores in distal femur fractures with the carbon fiber lateral plate or the nail plate combination as assessed by standard of care with VAS Pain scores. | 1 year
  Visual Analogue Scale (VAS) pain scores will be collected through standard of care at follow up visits at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year and the average for both treatment groups will be reported.
The average scores of the patient reported outcomes for the PROMIS PF in distal femur fractures with the carbon fiber lateral plate or the nail plate combination as assessed by standard of care patient reported outcome measures. | 1 year
  Patient-Reported Outcomes Measurement Information System Physical Function (PROMIS PF) scores will be collected through standard of care at follow up visits at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year and the average for both treatment groups will be reported.
The average scores of the patient reported outcomes for the PROMIS PI in distal femur fractures with the carbon fiber lateral plate or the nail plate combination as assessed by standard of care patient reported outcome measures. | 1 year
  Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS PI) scores will be collected through standard of care at follow up visits at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year and the average for both treatment groups will be reported.
The total number of patients with infection in the lateral plate versus the nail plate combination cohorts as assessed by standard of care wound check at follow up visits at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year. | 1 year
The average time to union (weeks) for the Carbo-fix lateral plate versus nail plate combination as assessed by standard of care radiographs | 1 year
The average time to return to activity (weeks) after the Carbo-fix lateral plate versus the nail plate combination as assessed by standard of care follow up visits at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year. | 1 year
The total number of patients undergoing reoperation with the Carbo-fix lateral plate versus the nail plate combination as assessed by standard of care follow up visits at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year. | 1 year
The total number of patients with malalignment of the femur with the Carbo-fix lateral plate versus the nail/plate combination as assessed by standard of care radiographs. | 1 year
The average surgical time (minutes) for patients in both treatment groups, as assessed by standard of care documentation. | 1 year
The average amount of blood loss (mL) for patients during surgical fixation for both treatment groups, as assessed by standard of care documentation. | 1 year
The average length of stay (days) for admission for surgical fixation for patients in each treatment group, as assessed by standard of care documentation. | 1 year
The total number of patients in each discharge disposition category (home, skilled nursing facility, or inpatient rehab) upon discharge after surgical fixation for each treatment group as assessed by standard of care documentation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Schweser, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

REFERENCES:
- [Background] Utility of Carbon Fiber Implants in Orthopedic Surgery: Literature Review Ronald Hillock, MD, Shain Howard, BS Reconstructive Review v. 4, n. 1 (31 March 2014): 55-55
- [Background] Garala K, Ramoutar D, Li J, Syed F, Arastu M, Ward J, Patil S. Distal femoral fractures: A comparison between single lateral plate fixation and a combined femoral nail and plate fixation. Injury. 2022 Feb;53(2):634-639. doi: 10.1016/j.injury.2021.11.011. Epub 2021 Nov 10. PMID 34836629
- [Background] Rodriguez EK, Boulton C, Weaver MJ, Herder LM, Morgan JH, Chacko AT, Appleton PT, Zurakowski D, Vrahas MS. Predictive factors of distal femoral fracture nonunion after lateral locked plating: a retrospective multicenter case-control study of 283 fractures. Injury. 2014 Mar;45(3):554-9. doi: 10.1016/j.injury.2013.10.042. Epub 2013 Nov 4. PMID 24275357
- [Background] Ebraheim NA, Martin A, Sochacki KR, Liu J. Nonunion of distal femoral fractures: a systematic review. Orthop Surg. 2013 Feb;5(1):46-50. doi: 10.1111/os.12017. PMID 23420747
- [Background] Khan AM, Tang QO, Spicer D. The Epidemiology of Adult Distal Femoral Shaft Fractures in a Central London Major Trauma Centre Over Five Years. Open Orthop J. 2017 Nov 13;11:1277-1291. doi: 10.2174/1874325001711011277. eCollection 2017. PMID 29290866